CLINICAL TRIAL: NCT04406571
Title: Reorganization of the Healthcare System During COVID-19 Pandemic: Impact on Management of Patients With Exocrine Pancreatic Cancer
Acronym: CAPANCOVID-19
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20042
Record Dates: First submitted 2020-05-27; First posted 2020-05-28 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: pancreatic adenocarcinoma; patient management; healthcare system reorganization; SARS-CoV-2
MeSH Terms: interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "pancreatic adenocarcinoma before COVID-19 containment " group: patients with pancreatic adenocarcinoma assessed during multidisciplinary meeting in one participating center between 01/09/2019 and 16/03/2020.
  Interventions: Other: Data record
- "pancreatic adenocarcinoma after COVID-19 containment " group: patients with pancreatic adenocarcinoma assessed during multidisciplinary meeting in one participating center between 17/03/2020 and 31/10/2020.
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record — Data record

SUMMARY:
Pancreatic adenocarcinoma will be the 2nd cause of death by cancer in Europe in 2030. Pancreatic adenocarcinoma has poor prognosis with an all-stages combined 5-year survival rate below 8%.

Since December 2019, a new coronavirus (Severe Acute Respiratory Syndrome Corona Virus 2, SARS-CoV-2) is responsible of COVID-19 infection with potentially severe respiratory syndrome or even multi-organ failure. An increased risk of severe COVID-19 infection in cancer patients is suggested in several Chinese series. Cancer care structures quickly reorganized to limit high-risk situations (diagnostic procedure, major surgery, cytotoxic poly-chemotherapy) and use alternatives such as on-hold chemotherapy. These reorganizations could be associated with a loss of chance for pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
The aim of this study is to study impact of reorganization of the healthcare system during COVID-19 pandemic on pancreatic adenocarcinoma patients management

ELIGIBILITY:
Inclusion criteria :

1. aged 18 or over,
2. with pancreatic adenocarcinoma diagnosed by anatomopathological specimen or without biopsy but with suspicion of pancreatic adenocarcinoma in presence of imaging techniques or Ca19.9 level without evidence for neuroendocrine tumor,
3. assessed during multidisciplinary meeting in one participating center between 01/09/2019 and 31/10/2020,
4. accepting to participate to the study,
5. with or without SARS-CoV-2 infection.

Exclusion criteria :

1. with neuroendocrine neoplasia
2. for whom histology showed non pancreatic
3. with cystadenoma or IPMN without invasive adenocarcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic adenocarcinoma diagnosed between 01/09/2019 and 31/10/2020.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Pancreatic adenocarcinoma treatment | 6 months
  curative surgery (with or without chemotherapy), chemotherapy only or exclusive supportive care

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Derived] Brugel M, Letrillart L, Evrard C, Thierry A, Tougeron D, El Amrani M, Piessen G, Truant S, Turpin A, d'Engremont C, Roth G, Hautefeuille V, Regimbeau JM, Williet N, Schwarz L, Di Fiore F, Borg C, Doussot A, Lambert A, Moulin V, Trelohan H, Bolliet M, Topolscki A, Ayav A, Lopez A, Botsen D, Piardi T, Carlier C, Bouche O. Impact of the COVID-19 pandemic on disease stage and treatment for patients with pancreatic adenocarcinoma: A French comprehensive multicentre ambispective observational cohort study (CAPANCOVID). Eur J Cancer. 2022 May;166:8-20. doi: 10.1016/j.ejca.2022.01.040. Epub 2022 Feb 10. PMID 35259629